CLINICAL TRIAL: NCT04140643
Title: Ozone Therapy as an Aid for Home Oral Hygiene. The Use of Aquolab in the Pregnant Woman.
Brief Title: Ozone Therapy for the Home Oral Hygiene of the Pregnant Woman.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Simona Tecco, Associate Professor, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EB2C
Record Dates: First submitted 2019-05-03; First posted 2019-10-28 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Pregnancy Gingivitis; Ozone
Keywords: Pregnancy; Oral Health; Ozone therapy; Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ozone therapy (Experimental): Oral hygiene instructions given by dental hygienist and home daily use of ozonated water delivering system.
  Interventions: Device: Ozonated water delivering device effects on the oral health of pregnant women
- Only oral hygiene instructions (Active Comparator): Oral hygiene instructions given by dental hygienist.
  Interventions: Behavioral: Oral hygiene instructions

INTERVENTIONS:
Device: Ozonated water delivering device effects on the oral health of pregnant women — Oral Hygiene instructions and use of an ozonated water delivering device in pregnant women for a period of 75 days.
  Arms: Ozone therapy
Behavioral: Oral hygiene instructions — Oral Hygiene instructions
  Arms: Only oral hygiene instructions

SUMMARY:
The aim of the present study is analyzing the effect of an domestic ozonated water delivering device on the oral health status of pregnant women.

Two groups of 30 women will be enrolled following a simple randomization scheme: the group A will be equipped with a domestic ozonated water delivering device and a control group B that will not be equipped with the device. The sample size was calculated with a power analysis performed starting from descriptive data differences obtained from a pilot study in order to achieve a power higher than 80 percent with an alpha error of 0.05 resulting in a minimum of 27 participants for each group.

The protocol was in accordance with the Declaration of Helsinki and was approved by the Ethical Committee of the IRCCS San Raffaele Hospital, all the participants will be informed about the aim of the study and will sign an informed consent form.

At the first examination (T0) the clinical oral hygiene parameters will be recorded on the enrolled participants of both the groups and they will be subjected to a professional oral hygiene procedure with appropriate home oral hygiene instructions. The same clinical oral hygiene parameters will be recorded also after 15 days (T1) and after 75 days (T2) from the first examination.

All the clinical procedures and data recording will be conducted by the operator X blind to the participants group while the operator Y will give the device and instruct the participants to its proper use.

After a descriptive analysis of the data, an analysis of the data distribution will be performed with the Kolmogorov-Smirnov test. According with the result of the data distribution analysis the differences between-groups and within-groups will be evaluated with the proper parametric or non-parametric test.

DETAILED DESCRIPTION:
The aim of the present study is analyzing the effect of an domestic ozonated water delivering device on the oral health status of pregnant women.

In the present study a total of 60 pregnant women will be recruited at the dental clinic of the IRCCS San Raffaele Hospital. These participants must adhere to the following inclusion criteria: legal age, pregnancy period between the 14 and 30 week, diagnosis positive for pregnancy gingivitis, presence of at least 20 teeth. The following exclusion criteria will be applied: absumption of alcohol during pregnancy, systemic diseases, chronic drug assumption, allergies, ongoing orthodontic therapies, positive periodontal screening recording (PSR).

The participants will be assigned to two groups following a simple randomization scheme: the group A will be equipped with a domestic ozonated water delivering device (Aquolab®, EB2C, Milan, Italy) and a control group B that will not be equipped with the device. The sample size was calculated with a power analysis performed starting from descriptive data differences obtained from a pilot study in order to achieve a power higher than 80 percent with an alpha error of 0.05 resulting in a minimum of 27 participants for each group. A total of 30 subjects will be assigned to each group in order to prevent possible drop-outs.

The protocol was in accordance with the Declaration of Helsinki and was approved by the Ethical Committee of the IRCCS San Raffaele Hospital, all the participants will be informed about the aim of the study and will sign an informed consent form.

At the first examination (T0) the clinical oral hygiene parameters will be recorded on the enrolled participants of both the groups and they will be subjected to a professional oral hygiene procedure with appropriate home oral hygiene instructions. The same clinical oral hygiene parameters will be recorded also after 15 days (T1) and after 75 days (T2) from the first examination.

All the clinical procedures and data recording will be conducted by the operator X blind to the participants group while the operator Y will give the device and instruct the participants to its proper use.

After a descriptive analysis of the data, an analysis of the data distribution will be performed with the Kolmogorov-Smirnov test. According with the result of the data distribution analysis the differences between-groups and within-groups will be evaluated with the proper parametric or non-parametric test.

ELIGIBILITY:
Inclusion Criteria:

* legal age
* pregnancy period between the 14 and 30 week
* diagnosis positive for pregnancy gingivitis
* presence of at least 20 teeth

Exclusion Criteria:

* absumption of alcohol during pregnancy
* systemic diseases
* chronic drug assumption
* allergies
* ongoing orthodontic therapies
* positive periodontal screening recording (PSR) at T1

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Periodontal Screening Recording (PSR) | 60 Days
  Code 0 - Colored area of probe remains completely visible in the deepest crevice in the sextant. No calculus or defective margins are detected. Gingival tissues are healthy with no bleeding after gentle probing.
  * Code 1 - Colored area of probe remains completely visible in the deepest probing depth in the sextant. No calculus or margins are detected. There is bleeding after gentle probing.
  * Code 2 - Colored area of probe remains completely visible in the deepest probing depth in the sextant. Supra- or subgingival calculus and/or defective margins are detected.
  Code 3 - Colored area of probe remains partly visible in the deepest probing depth in the sextant.
  • Code 4 - Colored area of probe completely disappears, indicating probing depth of greater than 5.5 mm.

SECONDARY OUTCOMES:
Bleeding of Probing (BOP) | 60 Days
  Expressed as Full Mouth Bleeding Score (FMPS), percentage of bleeding sites on the total number of available sites.
Plaque Index (PI) | 60 Days
  Expressed as Full Mouth Plaque Score (FMPS), percentage of plaque containing dental surfaces on the total number of available surfaces.
Probing Depth (PD) | 60 Days

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Gherlone, MD, MS, Study Chair — IRCCS San Raffaele Hospital
Locations (1):
- Dental Clinic, IRCCS San Raffaele Hospital, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Geisinger ML, Geurs NC, Bain JL, Kaur M, Vassilopoulos PJ, Cliver SP, Hauth JC, Reddy MS. Oral health education and therapy reduces gingivitis during pregnancy. J Clin Periodontol. 2014 Feb;41(2):141-8. doi: 10.1111/jcpe.12188. Epub 2013 Nov 19. PMID 24164645
- [Background] Jiang H, Xiong X, Buekens P, Su Y, Qian X. Use of mouth rinse during pregnancy to improve birth and neonatal outcomes: a randomized controlled trial. BMC Pregnancy Childbirth. 2015 Nov 25;15:311. doi: 10.1186/s12884-015-0761-3. PMID 26608342
- [Background] Villa A, Abati S, Pileri P, Calabrese S, Capobianco G, Strohmenger L, Ottolenghi L, Cetin I, Campus GG. Oral health and oral diseases in pregnancy: a multicentre survey of Italian postpartum women. Aust Dent J. 2013 Jun;58(2):224-9. doi: 10.1111/adj.12058. Epub 2013 May 5. PMID 23713644
- [Background] Almerich-Silla JM, Alminana-Pastor PJ, Boronat-Catala M, Bellot-Arcis C, Montiel-Company JM. Socioeconomic factors and severity of periodontal disease in adults (35-44 years). A cross sectional study. J Clin Exp Dent. 2017 Aug 1;9(8):e988-e994. doi: 10.4317/jced.54033. eCollection 2017 Aug. PMID 28936289
- [Derived] Tecco S, Nota A, D'Amicantonio T, Pittari L, Monti M, Polizzi E. Effects of an Ozonated Water Irrigator on the Plaque Index and Bleeding Index of Pregnant Women. J Clin Med. 2022 Jul 15;11(14):4107. doi: 10.3390/jcm11144107. PMID 35887871